CLINICAL TRIAL: NCT04834401
Title: Evaluating the Effect of Disease Modifying Therapy on Antibody Response to COVID19 Vaccination in People With Multiple Sclerosis
Brief Title: Effect of Disease Modifying Therapy on Antibody Response to COVID19 Vaccination in Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: St. Barnabas Medical Center (Other)
Responsible Party: Principal Investigator, Matthew A. Tremblay, Director of Multiple Sclerosis Research, St. Barnabas Medical Center
Other Study IDs: US-TYS-11909
Record Dates: First submitted 2021-04-02; First posted 2021-04-08 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Multiple Sclerosis; Covid19
Keywords: mRNA vaccine; Ocrelizumab; Natalizumab; Dimethyl Fumarate; Diroximel Fumarate; Interferon Beta; SARS-CoV-2
MeSH Terms: conditions — Multiple Sclerosis; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum will be stored for up to 2 years from enrollment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Natalizumab: Natalizumab (minimum of 6 doses at standard interval)
- Fumarates: Fumarates (dimethyl fumarate or diroximel fumarate)
- Interferon Beta 1a: Interferon Beta 1a (or pegylated Interferon Beta-1a)
- Ocrelizumab: Ocrelizumab (minimum of 2 full cycles of 600mg)

SUMMARY:
This observational study is intended to evaluate the effect of disease modifying therapies on antibody responses to the mRNA-1273 vaccine (Moderna) for COVID-19. We hypothesize that the use of certain disease modifying therapies, particularly ocrelizumab, will mute and/or shorten the duration of humoral response to mRNA vaccines.

DETAILED DESCRIPTION:
COVID-19 is a potentially fatal respiratory illness, caused by the novel coronavirus, SARS-CoV-2, which developed into a pandemic claiming the lives of over 500,000 people in the United States and over 2.5 million worldwide. Antibodies against the spike glycoprotein are believed to confer immunity to SARS-CoV-2. Multiple sclerosis (MS) is an autoimmune disease of the central nervous system, which is typically treated with immunomodulating medications, referred to as disease modifying therapies (DMTs). Some DMTs resulted in a diminished capacity to develop antibodies against natural infection with SARS-CoV-2. This study is designed to evaluate and compare the effect of DMTs on antibody response to mRNA vaccines for COVID-19. Serum samples will be collected from 30 participants per treatment arm at 8 weeks, 24 weeks, 36 weeks, and 48 weeks, following vaccination with mRNA-1273. Geometric mean titers of anti-SARS-CoV-2 spike IgG will be measured to evaluate and compare peak antibody titers, as well as the duration of antibody response. The results will likely impact clinical decision-making, and guide treatment strategies for safely managing MS during the ongoing pandemic.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18 to 65 years inclusive
2. Patients who have signed written informed consent.
3. Patients stable on current MS DMT for >6 months including:

   * Natalizumab (received a minimum of 6 doses per USPI)
   * Fumarates (dimethyl fumarate or diroximel fumarate)
   * Interferon Beta 1a (or pegylated Interferon Beta-1a)
   * Ocrelizumab (received a minimum of 2 full cycles per USPI)

Exclusion Criteria:

1. Known history of SARS-CoV-2 infection
2. Is pregnant or breastfeeding
3. ≤6 months on current therapy (MS Participants)
4. Participation in another investigational study
5. Recent immunization with a non-COVID vaccine (within 4 weeks)
6. Known or suspected allergy or history of anaphylaxis or other significant adverse reaction to the COVID-19 vaccine or its excipients
7. Absolute lymphocyte count <0.5 x 10^9/L
8. Concurrent Intravenous or Subcutaneous Immunoglobulin treatment (IVIG/SCIG)
9. Received systemic corticosteroids < 30 days prior to Vaccine Dose 1

Visit and Assessment Schedule:

Participants will agree to five visits during the study and serum will be collected at the following time points:

* Baseline/Screening visit
* 8 weeks after 1st dose/4 weeks after 2nd dose (+/- 1 week)
* 24 weeks (+/- 2 weeks)
* 36 weeks (+/- 4 weeks)
* 48 weeks (+/- 4 weeks)

Approximately 20ml of blood will be collected per patient per each visit.

Data Collection Plan and Patient Privacy Protection Prior to any testing under this protocol, including screening tests and assessments, candidates must also provide all authorizations required by local law (e.g., PHI authorization in North America).

The subject will not be identified by name in the CRF or in any study reports, and these reports will be used for research purposes only. Ethics committees and various government health agencies may inspect the records of this study. Every effort will be made to keep the subject's personal medical data confidential.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants will be identified from the MS Center utilizing the electronic medical record, clinic visits or telephone encounters related to COVID-19 vaccination and recruited consecutively. Patients who appear to meet eligibility criteria will be contacted by research staff and offered informed consent using the Multiple Sclerosis Comprehensive Care Center standard protocol. If possible the baseline serum sample will be collected at the initial research visit, following the informed consent process.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-05-17 (Actual)

PRIMARY OUTCOMES:
Geometric mean titers (GMT) of anti-SARS-CoV-2 spike IgG for each treatment at 8 weeks from initial vaccination dose | 8 weeks
  Serum Sample

SECONDARY OUTCOMES:
Proportion of participants with >4 fold increase in anti-SARS-CoV-2 spike IgG between baseline and 8 weeks | 8 weeks
  Serum sample
Proportion of participants with >2 fold increase in anti-SARS-CoV-2 spike IgG between baseline and 8 weeks | 8 weeks
  Serum Sample
Median time from peak to complete absence of anti-SARS-CoV-2 IgG for each treatment arm | 18 months
  Serum Sample
Proportion of spike-specific T-cells/Total T cells | 36 Weeks
  Whole Blood Sample

OTHER OUTCOMES:
Proportion of participants with known vaccine-related side effects | 8 weeks
  Questionnaire
COVID-19 Infections | 18 months
  Number of participants with PCR-confirmed COVID-19 infection following vaccination
Effect of Duration of DMT use on Humoral Response to mRNA-1273 | 8 week
  Correlation between duration of DMT and GMT values for SARS-CoV-2 IgG within each treatment arm

CONTACTS AND LOCATIONS:
Overall Officials: Matthew A Tremblay, MD, PhD, Principal Investigator — RWJBarnabas Health
Locations (1):
- Saint Barnabas Medical Center, Livingston, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided